CLINICAL TRIAL: NCT04422899
Title: A Phase I Study of the Safety, Pharmacokinetics, and Duration of Effect of Intravitreally Administered AIV007 Gel Suspension in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: Effect of Intravitreally Administered AIV007 in Subjects With Neovascular Age-Related Macular Degeneration
Acronym: nAMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AiViva BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AIV007-E01
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AIV007 Treatment Dose 1 (Experimental): Intravitreal, Dose 1
  Interventions: Drug: AIV007
- AIV007 Treatment Dose 2 (Experimental): Intravitreal, Dose 2
  Interventions: Drug: AIV007
- AIV007 Treatment Dose 3 (Experimental): Intravitreal, Dose 3
  Interventions: Drug: AIV007

INTERVENTIONS:
Drug: AIV007 — intravitreal

SUMMARY:
To determine safety, pharmacokinetics, and duration of effect of intravitreally administered AIV007 gel suspension in subjects with neovascular age-related macular degeneration

DETAILED DESCRIPTION:
AIV007 is a multiple kinase inhibitor of vascular endothelial growth factor receptors (VEGFR 1, -2 & -3); fibroblast growth factor receptors (FGFR-1, -2, -3 & -4); and platelet-derived growth factor receptors (PDGFR-α & β)1. Lenvatinib is the active pharmaceutical ingredient in AIV007 formulation that is FDA-approved for oral administration for patients with advanced renal cell carcinoma (RCC), differentiated thyroid cancer (DTC), unresectable hepatocellular carcinoma (HCC), and advanced endometrial carcinoma (Lenvima USPI 2021; NDA 206947). AIV007 is a novel, thermoresponsive gel suspension for intravitreal administration proposed to form a durable depot inside the eye. This monotherapy is being evaluated for the treatment of retinal and choroidal vascular disease. A single intravitreal treatment in 3 subjects was evaluated using 2 doses to evaluate depot formation, safety and biological activity by measuring visual acuity, reduction in retinal fluids associated with vision and effects of fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 50 years
2. Subjects must provide written informed consent before any study-related procedures are performed
3. Active subfoveal CNV in the study eye secondary to AMD that has previously been treated with at least 3 intravitreal injections of an anti-VEGF agent
4. BCVA in the study eye

   1. Sentinel subjects only: 65 ETDRS letters (20/50 Snellen equivalent) or worse
   2. All other subjects: 78 to 35 ETDRS letters (20/32 to 20/200 Snellen equivalent)
5. Clear ocular media and adequate pupil dilation in both eyes to permit good quality photographic imaging

Exclusion Criteria:

1. Previous treatment for nAMD in the study eye, other than standard-of-care anti- VEGF IVT injection, eg, cell therapy, brachytherapy, gene therapy
2. Treatment with anti-VEGF in the non-study eye 2 weeks prior to baseline
3. Presence of diabetic retinopathy or glaucoma in either eye
4. Spherical equivalent for refractive error in the study eye of worse than 8.0 diopters of myopia (prior to cataract or refractive surgery)
5. Presence of active infection or inflammation within 30 days prior to screening
6. Presence of contraindications to anti-VEGF treatment, including myocardial infarction, any cardiac event requiring hospitalization, treatment for acute congestive heart failure, transient ischemic attack, or stroke within the last 3 months of baseline
7. Uncontrolled hypertension or diabetes mellitus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events | approximately 224 days
  Incidence of adverse events

SECONDARY OUTCOMES:
Mean change from baseline in BCVA | approximately 224 days
  Number of ETDRS letters
Mean change from baseline in central subfield thickness as measured by optical coherence tomography | approximately 224 days
  OCT read by a central reading center
Mean time to rescue medication (administration of anti-VEGF medication) | approximately 224 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Salehi Retina Institute, Huntington Beach, California
  - Retina Research Institute of Texas, Abilene, Texas